CLINICAL TRIAL: NCT00135473
Title: Prospective Randomized Multicenter Study on the Influence of Colloid vs Crystalloid Volume Resuscitation and of Intensive vs Conventional Insulin Therapy on Outcome in Patients With Severe Sepsis and Septic Shock
Brief Title: Efficacy of Volume Substitution and Insulin Therapy in Severe Sepsis (VISEP Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SepNet - Critical Care Trials Group (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); B. Braun Melsungen AG (Industry); Novo Nordisk A/S (Industry); HemoCue (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SEPNET-200304; 01 KI 0106 (BMBF)
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Severe sepsis; septic shock; volume substitution; intensive insulin therapy; colloids; crystalloids; outcome; safety
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Hydroxyethyl Starch Derivatives; sterofundin; Insulin

INTERVENTIONS:
Drug: 10% Hemohes® (10% Hydroxyethyl starch)
Drug: Sterofundin® (Ringer lactate solution)
Drug: Actrapid® (Insulin)

SUMMARY:
The purpose of this trial is to determine the influence of colloid versus crystalloid volume resuscitation and of intensive vs conventional insulin therapy on morbidity and mortality of patients with severe sepsis and septic shock.

DETAILED DESCRIPTION:
Severe sepsis and septic shock have a high mortality. Research has concentrated on adjunctive sepsis therapies; the role of supportive measures is comparatively unclear. In Europe the use of colloids is widespread, but there is no evidence on the role of either crystalloid or colloid volume therapy in sepsis. Recently, a higher incidence of kidney failure in sepsis was reported after administration of colloids.

In critical illness, a significant reduction in mortality was recently achieved by strict glycemic control, however it has to be determined whether this is true and safe for patients with sepsis as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the criteria of "severe sepsis" or "septic shock" according to the Society of Critical Care Medicine/American College of Chest Physicians (SCCM/ACCP) definitions not longer than 24 hours before ICU admission or 12 hours after ICU admission

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Known allergy against hydroxyethyl starch
* Pre-treatment with > 1000ml hydroxyethyl starch within 24 hours before inclusion
* Pre-existing kidney failure requiring dialysis or serum creatinine value > 320 mmol/l (3,6 mg/dl)
* Intracerebral hemorrhage
* Severe head trauma with edema
* FiO2 at time of study inclusion > 0,7
* Heart failure (New York Heart Association [NYHA] IV)
* Enrolment in another interventional study
* Immune suppression (cytostatic chemotherapy, steroid therapy, AIDS)
* Do not resuscitate (DNR) order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2003-04; Study Completion 2005-09

PRIMARY OUTCOMES:
Mortality (28 day)
Morbidity (mean sepsis-related organ failure assessment [SOFA] score during intensive care unit length of stay [ICU LOS])

SECONDARY OUTCOMES:
Frequency of acute kidney failure
Time until hemodynamic stabilization
Frequency of therapy with vasopressors (in days)
Course of SOFA sub-scores
Frequency of hemorrhages under hydroxyethyl starch (HES) therapy
Frequency of hypoglycemia under intensive insulin therapy
Frequency of critical illness polyneuropathy (CIP)
90 day Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Reinhart, MD, Study Chair — F.-Schiller-University Jena, Germany; Thomas Deufel, MD, Study Director — F.-Schiller-University Jena, Germany; Markus Löffler, MD, Study Director — University of Leipzig
Locations (16):
- Germany (16):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - VIVANTES Klinikum Neukölln II, Berlin
  - Charité I Campus Virchow-Klinikum, Berlin
  - Städtisches Klinikum Brandenburg GmbH, Brandenburg
  - Krankenhaus Dresden Friedrichstadt, Dresden
  - Universität Carl-Gustav-Carus, Dresden
  - HELIOS Klinikum Erfurt, Erfurt
  - Universität Erlangen-Nürnberg, Erlangen
  - Georg-August-Universität Göttingen, Göttingen
  - Ernst-Moritz-Arndt-Universität, Greifswald
  - Martin-Luther-Universität Halle/Wittenberg, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig

REFERENCES:
- [Derived] Brunkhorst FM, Engel C, Bloos F, Meier-Hellmann A, Ragaller M, Weiler N, Moerer O, Gruendling M, Oppert M, Grond S, Olthoff D, Jaschinski U, John S, Rossaint R, Welte T, Schaefer M, Kern P, Kuhnt E, Kiehntopf M, Hartog C, Natanson C, Loeffler M, Reinhart K; German Competence Network Sepsis (SepNet). Intensive insulin therapy and pentastarch resuscitation in severe sepsis. N Engl J Med. 2008 Jan 10;358(2):125-39. doi: 10.1056/NEJMoa070716. PMID 18184958